CLINICAL TRIAL: NCT06412692
Title: The Effect of Motivational Interviewıng Technique on Social Anxiety and Quality of Life of Adolescents With Epilepsy
Brief Title: Motivational Interviewing in Adolescents With Epilepsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, ELİZ GECTAN, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: İzmirKCU-GECTAN-001
Record Dates: First submitted 2024-04-30; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Pediatric ALL
Keywords: Epilepsy; Adolescent; Motivational Interviewing
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Epilepsy

STUDY DESIGN:
Intervention Model Description: In our study; The motivational interview technique will be applied to the intervention group individually by the researcher at 2-week intervals, including a preliminary interview and 6 motivational interview sessions.
Who Masked: Outcomes Assessor
Masking Description: Randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Motivational Interviewing Technique (Experimental): The Motivational Interviewing Technique Group (n=36) An equal number of patients will be classified by gender. Before the interview, each adolescent: Informed Consent Form, Personal Information Form, Social Anxiety Scale for Adolescents, Children's General Quality of Life Scale, and KINDL Epilepsy Quality of Life Module for Children will be applied. Interviews will be held in the training room next to the Child Neurology Polyclinic. In our study; The motivational interviewing technique will be applied to the experimental group individually by the researcher at 2-week intervals, including a preliminary interview and 6 motivational interview sessions. Each motivational interview will last approximately 40-50 minutes. One day before the motivational interview day, the experimental group will be informed by calling their registered phone numbers. The surveys will be re-administered after the end of the interview sessions. Surveys will be administered again after 1 month.
  Interventions: Other: The Motivational Interviewing Technique
- No Intervention (No Intervention): No Intervention Group (n=36) Equal numbers of patients will be stratified according to gender. Adolescents without intervention; Patient Consent Form, Personal Information Form, Social Anxiety Scale in Adolescents, Child's General Quality of Life Scale, KINDL Epilepsy Quality of Life Module in Children will be applied. Routine follow-up and treatment will continue. The duration of the pre-interview and 6 motivational interviews will be calculated and the scales will be applied again.The surveys will be administered again after 1 month.

INTERVENTIONS:
Other: The Motivational Interviewing Technique — Motivational interviewing technique applied to adolescents with epilepsy; It is thought that it will be effective in reducing social anxiety and increasing the quality of life of adolesce.
  Arms: The Motivational Interviewing Technique

SUMMARY:
Epilepsy is the most common serious neurodevelopmental disorder of childhood characterized by recurrent seizures, affecting approximately 0.9% of children and adolescents worldwide. Although epileptic seizures are an important element of epilepsy in children, there are many neurological, mental health and cognitive comorbidities in childhood epilepsy that increase the burden of the disease and cause a decrease in quality of life. Motivational interviewing has been found to have a positive effect on the treatment and prevention of chronic diseases; It is a patient-centered counseling that explores, strengthens, and directs the individual's motivation for change.

DETAILED DESCRIPTION:
Adolescence period; It is an important stage of development in which the self-concept develops, self-related schemas are created and carried into adulthood. During this formative period of life; Adolescents experience increasing levels of uncertainty and self-consciousness as they progress through the task of identity formation. It is greatly influenced by social interactions, especially interactions with peers.Children and adolescents with epilepsy are at increased risk for social problems, reduced social competence, poor social skills, and deficits in social communication compared to healthy children. Compared to youth with other chronic diseases, youth with epilepsy have higher rates of comorbid neurological disorders, academic failure, poor social skills, stigma, poor quality of life, and behavioral health problems (e.g., anxiety, depression). They often experience low quality of life because they feel unsafe and fear having a seizure in public. In a study aiming to investigate the factors affecting the level of social anxiety in epilepsy, it was concluded that social anxiety is independently associated with low quality of life. In a meta-analysis study; It was concluded that the motivational interviewing method applied by nurses increased the quality of life of individuals with chronic diseases. When the literature was examined, no study was found that addressed the motivational interviewing technique applied to the social anxiety and quality of life of adolescents with epilepsy. Motivational Interviewing Technique applied to adolescents with epilepsy; It is thought that it will be effective in reducing social anxiety and increasing the quality of life by enabling adolescents to become aware of their situation, get rid of the ambivalent (opposite emotional state) they experience, and take action to change.

ELIGIBILITY:
Inclusion Criteria:

* Be between the ages of 12-15
* Having epilepsy for at least six months
* Having a high score on the Social Anxiety Scale for Adolescents
* Having a low score on the General Child Life Quality Scale
* Low scores on the KINDL Epilepsy Quality of Life Module for Children
* No mental disability
* Able to communicate (can speak and understand Turkish, has no speech disorder)
* Being literate
* Not having any other chronic disease
* Being willing to participate in the study

Exclusion Criteria:

-Not attending at least one of the interviewing

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — Experimental and control groups were selected based on randomization gender.
Enrollment: 72 (Estimated)
Dates: Start 2023-11-18 (Actual); Primary Completion 2024-05-20 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
"Social Anxiety Scale for Adolescents" [Time Frame: After the motivational interviewing technique] | 3 months
  A high score on the Social Anxiety Scale for Adolescents indicates high anxiety.
''KINDL Epilepsy Quality of Life Module for Children'' [Time Frame: After the motivational interviewing technique] | 3 months
  A high score on the KINDL Epilepsy Quality of Life Module for Children indicates good healthy quality of life.
"Children's General Quality of Life Scale'' [Time Frame: After the motivational interviewing technique] | 3 months
  A high score on the Children's General Quality of Life Scale for Children indicates good healthy quality of life.
"Social Anxiety Scale for Adolescents" [Time Frame: 1 month after the Motivational Interviewing Technique] | 1 months
  A high score on the Social Anxiety Scale for Adolescents indicates high anxiety.
''KINDL Epilepsy Quality of Life Module for Children'' [Time Frame: 1 month after the Motivational Interviewing Technique] | 1 months
  A high score on the KINDL Epilepsy Quality of Life Module for Children indicates good healthy quality of life.
"Children's General Quality of Life Scale" [Time Frame: 1 month after the Motivational Interviewing Technique] | 1 months
  A high score on the Children's General Quality of Life Scale for Children indicates good healthy quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- İzmirKCU, Izmir, Çigli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Clifford LM, Brothers SL, Lang A. Self-Disclosure Patterns Among Children and Youth with Epilepsy: Impact of Perceived-Stigma. Adolesc Health Med Ther. 2023 Feb 5;14:27-43. doi: 10.2147/AHMT.S336124. eCollection 2023. PMID 36776152
- [Background] Tolchin B, Baslet G, Martino S, Suzuki J, Blumenfeld H, Hirsch LJ, Altalib H, Dworetzky BA. Motivational Interviewing Techniques to Improve Psychotherapy Adherence and Outcomes for Patients With Psychogenic Nonepileptic Seizures. J Neuropsychiatry Clin Neurosci. 2020 Spring;32(2):125-131. doi: 10.1176/appi.neuropsych.19020045. Epub 2019 Aug 30. PMID 31466516
- [Background] Tolchin B, Baslet G, Suzuki J, Martino S, Blumenfeld H, Hirsch LJ, Altalib H, Dworetzky BA. Randomized controlled trial of motivational interviewing for psychogenic nonepileptic seizures. Epilepsia. 2019 May;60(5):986-995. doi: 10.1111/epi.14728. Epub 2019 Apr 13. PMID 30980679
- [Background] Vallabhan MK, Jimenez EY, Nash JL, Gonzales-Pacheco D, Coakley KE, Noe SR, DeBlieck CJ, Summers LC, Feldstein-Ewing SW, Kong AS. Motivational Interviewing to Treat Adolescents With Obesity: A Meta-analysis. Pediatrics. 2018 Nov;142(5):e20180733. doi: 10.1542/peds.2018-0733. Epub 2018 Oct 22. PMID 30348753
- [Background] Aburahma SK, Hammouri H, Hazaimeh E, Jbarah O, Nassar A, Almasri A, Al Momani M, Bashtawi M. Social impairment in children with epilepsy assessed by the social responsiveness scale. Clin Child Psychol Psychiatry. 2021 Oct;26(4):1170-1181. doi: 10.1177/13591045211033176. Epub 2021 Jul 16. PMID 34271834
- [Background] Hosseini N, Mokhtari S, Momeni E, Vossoughi M, Barekatian M. Effect of motivational interviewing on quality of life in patients with epilepsy. Epilepsy Behav. 2016 Feb;55:70-4. doi: 10.1016/j.yebeh.2015.10.012. Epub 2016 Jan 12. PMID 26773672
- [Background] Lu Y, Zhong R, Li M, Zhao Q, Zhang X, Hu B, Lin W. Social anxiety is associated with poor quality of life in adults with epilepsy in Northeast China: A cross-sectional study. Epilepsy Behav. 2021 Apr;117:107866. doi: 10.1016/j.yebeh.2021.107866. Epub 2021 Mar 5. PMID 33684784
- [Background] Uzun S, Ozmaya E. The effect of motivational interview conducted by nurses on quality of life: Meta-analysis. Perspect Psychiatr Care. 2022 Oct;58(4):2449-2459. doi: 10.1111/ppc.13080. Epub 2022 Apr 5. PMID 35383938